CLINICAL TRIAL: NCT03871673
Title: A Novel Approach to Treatment of Hepatic Glycogen Storage Diseases: a Study Based on the Use of Uncooked Sweet Manioc Starch
Brief Title: The Use of Uncooked Sweet Manioc Starch to Treat Hepatic Glycogen Storage Diseases
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Collaborators: Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government); Fundação Médica do Rio Grande do Sul (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 160056
Record Dates: First submitted 2019-03-09; First posted 2019-03-12 (Actual); Last update posted 2023-09-26 (Actual); Status verified 2023-09

CONDITIONS: Glycogen Storage Disease Type I
Keywords: Hepatic Glycogen Storage Diseases; Treatment; Clinical trial; Cornstarch; Sweet manioc starch
MeSH Terms: conditions — Glycogen Storage Disease Type I | interventions — Starch

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cornstarch (Active Comparator): Ingestion of cornstarch, the standard treatment for hepatic Glycogen Storage Diseases.
  Interventions: Dietary Supplement: Cornstarch
- Sweet manioc starch (Experimental): Ingestion of sweet manioc starch, the starch in study.
  Interventions: Dietary Supplement: Sweet manioc starch

INTERVENTIONS:
Dietary Supplement: Sweet manioc starch — 100 g of starch diluted in 200 ml of water at room temperature In the subsequent night the patient is crossed over to the other starch.
  Arms: Sweet manioc starch
Dietary Supplement: Cornstarch — 100 g of starch diluted in 200 ml of water at room temperature In the subsequent night the patient is crossed over to the other starch.
  Arms: Cornstarch

SUMMARY:
Hepatic Glycogen Storage Diseases are a group of 10 serious genetic diseases that present in childhood and are characterized more frequently by the occurrence of repetitive hypoglycemia and dyslipidemia. Regarding treatment, the most commonly used strategy is the frequent administration of uncooked cornstarch, in average, every 4 hours. Although this treatment is successful, the use of large amounts of cornstarch can lead to overweight and, especially, to the decrease in the quality of life of patients and caregivers, due to the need to use the starch during the night. The search for a treatment that is widely available and that can lead to the prolongation of the fasting time, can collaborate to improve the care of these patients. The main scientific question to be answered by this research is: does sweet manioc starch, a Brazilian product, safely prolong the fasting time (with normoglycemia) of the patients as already suggested in experimental models? Main objective: To evaluate the efficacy and safety of the use of uncooked Sweet Manioc Starch in the treatment of patients with hepatic Glycogen Storage Diseases, using as model the Glycogen Storage Diseases type Ia.

DETAILED DESCRIPTION:
A randomize and crossover study will be conducted on two consecutive days, comparing the use of classic cornstarch to the use of sweet manioc starch in patients with Glycogen Storage Disease type Ia. Ten patients diagnosed with Glycogen Storage Disease type Ia, confirmed by genetic analysis, will be included in the study. Sweet manioc starch and cornstarch, both of Brazilian origin, were analyzed in a previous study of the team in the artificial gastrointestinal model (TIM-1). They will be supplied uncooked, in the same way that cornstarch is currently used in the treatment of hepatic Glycogen Storage Diseases. Doses administered to patients will be 100 g of starch diluted in 200 ml of water at room temperature. To carry out the study, the patients will remain two consecutive nights in the hospital. They will remain in their normal diet until the administration of the starches at 22 hours. To perform the test, at 10 pm blood collection will be performed and after that the patient will ingest the starch (cornstarch or sweet manioc starch, determined by previous randomization). In sequence, blood collection will be performed every hour until the patient has a serum glucose value below 70mg/dL or after the patient stays 10h in a fast. Afterwards, the patient will return to his usual diet until the next test at 22 hours. The same procedures will be performed on the second night, the only change will be the starch used, and if the patient ingested uncooked cornstarch the first night, the same night will ingest the sweet manioc starch, or the opposite.If the patient has hypoglycaemia during the study, it will be discontinued.

ELIGIBILITY:
Inclusion Criteria:

* patients with a confirmed molecular diagnosis of glycogen storage disease type Ia who are already on uncooked cornstarch therapy

Exclusion Criteria:

-

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2017-04-29 (Actual); Primary Completion 2019-08-30 (Actual); Study Completion 2021-05-31 (Actual)

PRIMARY OUTCOMES:
Duration of normoglycemia | up to 10 hours
  To verify the normoglycemia will be accessed glucose level. The glucose dosage will be performed by hexokinase enzyme assay. Peripheral blood samples will be collected to determine the baseline value and every hour.

SECONDARY OUTCOMES:
Glucose levels | up to 10 hours
  The glucose dosage will be performed by hexokinase enzyme assay. Peripheral blood samples will be collected to determine the baseline value and every hour.
Lactate levels | up to 10 hours
  The lactase dosage will be performed by colorimetric (Lactate → Pyruvate). Peripheral blood samples will be collected to determine the baseline value and every hour.
Insulin levels | up to 10 hours
  The insulin dosage will be performed by microparticle chemiluminescent immunoassay. Peripheral blood samples will be collected to determine the baseline value and every hour.

CONTACTS AND LOCATIONS:
Overall Officials: Ida D Schwartz, Dr, Principal Investigator — Hospital de Clínicas de Porto Alegre
Locations (1):
- Ida Vanessa D Schwartz, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Monteiro VCL, de Oliveira BM, Dos Santos BB, Sperb-Ludwig F, Refosco LF, Nalin T, Derks TGJ, Moura de Souza CF, Schwartz IVD. A triple-blinded crossover study to evaluate the short-term safety of sweet manioc starch for the treatment of glycogen storage disease type Ia. Orphanet J Rare Dis. 2021 Jun 3;16(1):254. doi: 10.1186/s13023-021-01877-3. PMID 34082801
- See also: A triple-blinded crossover study to evaluate the short-term safety of sweet manioc starch for the treatment of glycogen storage disease type Ia — https://pubmed.ncbi.nlm.nih.gov/34082801/